CLINICAL TRIAL: NCT01260064
Title: The Outcomes of Various Appendectomy Techniques in a High-volume Center.
Brief Title: Open Appendectomy Versus Laparoscopic Appendectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bakirkoy Dr. Sadi Konuk Research and Training Hospital (Other Government)
Responsible Party: General Surgery Clinics, Dr. Sadi Konuk Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Frumious
Record Dates: First submitted 2010-12-13; First posted 2010-12-15 (Estimated); Last update posted 2011-05-26 (Estimated); Status verified 2011-05

CONDITIONS: Appendicitis
Keywords: Appendicitis; Open appendectomy; Laparoscopic appendectomy; Endoclip; Intracorporeal suture; Quality-of-life
MeSH Terms: conditions — Appendicitis | interventions — Open Abdomen Techniques

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Open appendectomy (Active Comparator): The subjects will have open appendectomy procedure.
  Interventions: Procedure: Open appendectomy
- Metal endoclip (Active Comparator): The subjects will have laparoscopic appendectomy in which the appendiceal stump is secured by metal endoclips.
  Interventions: Procedure: Laparoscopic appendectomy with metal endoclips
- Intracorporeal suture ligation (Active Comparator): The subjects will have laparoscopic appendectomy in which the appendiceal stump is secured by intracorporeal suture ligation.
  Interventions: Procedure: Laparoscopic appendectomy with suture ligation

INTERVENTIONS:
Procedure: Open appendectomy — The subjects will have traditional open appendectomy procedure.
  Other Names: Open technique
  Arms: Open appendectomy
Procedure: Laparoscopic appendectomy with metal endoclips — The subjects will have laparoscopic appendectomy in which the appendiceal stump is secured by metal endoclips.
  Other Names: Metal endoclip
  Arms: Metal endoclip
Procedure: Laparoscopic appendectomy with suture ligation — The subjects will have laparoscopic appendectomy in which the appendiceal stump is secured by intracorporeal suture ligation.
  Other Names: Intracorporeal suture ligation
  Arms: Intracorporeal suture ligation

SUMMARY:
1. Laparoscopic appendectomy may not be a superior procedure when compared with open appendectomy; 2. Various modifications in laparoscopic appendectomy procedure may reduce the technical diffuculty and overall costs.

DETAILED DESCRIPTION:
The study will be a prospective randomized clinical trial. Totally 150 patients who are diagnosed to have acute appendicitis will be randomly divided into 3 equal groups (n=50 for each group). First group will have traditional open appendectomy procedure; second group will have laparoscopic appendectomy procedure in which appendiceal stump is secured by metal endoclips; and third group will have laparoscopic appendectomy procedure in which appendiceal stump is secured by intracorporeal suture ligation. The preoperative parameters that will be obtained for all patients are: detailed information for communication, patient history, age, gender, the presence of spesific symptoms (nausea, vomiting, loss of appetite, right lower quadrant pain), the presence of clinical signs, laboratory findings, and radiological findings. The peroperative parameters that will be recorded are: operative time, the type and the length of incisions, the number of trocars, operative findings, details of laparoscopic technique, generic name of prophylactic antibiotic, and the presence of additional findings. All of the patients will undergo a clinical evaluation by attending surgeon on the 5th, the 15th, and the 30th postoperative day. The postoperative clinical evaluation will include the examination of the patient for surgical site infection and other wound complications, and the performance of a spesific quality-of-life index questionnaire. In the end of the study, all parameters and quality-of-life scores will undergo statistical analysis.

ELIGIBILITY:
Inclusion Criteria:

* The patients with a preoperative diagnosis of acute appendicitis

Exclusion Criteria:

* The patients who are not volunteered to join the study
* The patients who are diagnosed to have peroperative or histopathological pathology other than acute appendicitis
* The patients who have additional pathologies accompanying acute appendicitis

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2010-10; Primary Completion 2011-04 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Quality of life. | 1 month
  Quality of life after various appendectomy procedures will be measured by a spesific quality-of-life index.

SECONDARY OUTCOMES:
Cost-effectivity | 1 month
  The study will reveal which procedure for appendectomy is the most cost-effective one.

CONTACTS AND LOCATIONS:
Overall Officials: Halil Alis, MD, Study Director — Dr. Sadi Konuk Training and Research Hospital
Locations (1):
- Dr. Sadi Konuk Training and Research Hospital, Istanbul, Turkey (Türkiye)